CLINICAL TRIAL: NCT05242458
Title: Real-world Evidence for the Effectiveness and Safety of Ustekinumab Treatment in Children With Crohn's Disease: A Retrospective Cohort Study Using the ImproveCareNow Registry Data
Brief Title: A Study of Ustekinumab Treatment in Children With Crohn's Disease
Acronym: REALITI
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: ImproveCareNow (ICN) (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: CR109167; CNTO1275CRD3010 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-02-15; First posted 2022-02-16 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Participants with Crohn's Disease (CD): Participants with moderate-to-severe active CD enrolled in ImproveCareNow (ICN) pediatric Inflammatory bowel disease (IBD) registry will be observed who are being treated with ustekinumab under real world setting and will be divided into 9 cohorts. Cohorts 1-6 for age group >=2 to <18 years (pediatric), cohorts 7-9 for young adults within age group >=18 to <26 years. Cohort 1: participants with moderate-severe CD and body weight >=40 kg, cohort 2: participants with moderate-severe CD and body weight <40 kg, cohort 3: all participants with moderate-severe CD, cohort 4: participants with active disease and body weight >=40 kg, cohort 5: participants with active disease and body weight <40 kg, cohort 6: all participants treated with ustekinumab, cohort 7: young adults with moderate-severe CD, cohort 8: young adults with active-disease; and cohort 9: all young adults treated with ustekinumab. Only data available per routine clinical practice will be collected within this study.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — No interventions will be administered as a part of this study. Participants will receive ustekinumab as per their routine clinical practice.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of ustekinumab in achieving clinical remission in pediatric participants (greater than or equal to [>=] 2 to less than [<] 18 years and weight >= 40 kilograms [kg] at baseline).

ELIGIBILITY:
Inclusion Criteria:

* Having at least one ICN visit with documented new use of ustekinumab
* Participants with a documented Crohn's disease (CD) diagnosis at the time ustekinumab was initiated (that is, Baseline); If diagnosis at baseline is missing, then the diagnosis from previous visit within study window will be utilized
* Having at least one ICN visit prior to the ICN visit when ustekinumab is first documented
* Having received first dose of ustekinumab on or before June 22, 2019
* Having provided informed consent for use of ICN data for research purposes

Exclusion Criteria:

* Documented exposure to ustekinumab before enrollment in ICN (by chart review)

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population includes pediatric participants (age greater than or equal to [>=] 2 to less than [<] 18 years with body weight >=40 kilograms [kg]) and young adults (age >= 18 to < 26 years) with moderately to severely active Crohn's disease. The primary study population will be pediatric participants who have moderate to severe disease activity defined as short pediatric Crohn's disease activity index (sPCDAI) >= 30, are treated with ustekinumab, and are followed at an ImproveCareNow (ICN) center.
Sampling Method: Non-Probability Sample
Enrollment: 545 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Cohort 1: Percentage of Pediatric Participants with Clinical Remission at Week 52 | Week 52
  Percentage of Pediatric participants with clinical remission at Week 52 will be reported. Clinical remission is defined by short pediatric Crohn's disease activity index (sPCDAI) less than or equal to (<=) 10.

SECONDARY OUTCOMES:
Cohort 7: Percentage of Young Adult Participants with Clinical Remission at Week 52 | Week 52
  Percentage of young adult participants with clinical remission at Week 52 will be reported.
Cohorts 2, 3, 4, 5, 6, 8 and 9: Percentage of Participants with Clinical Remission at Week 52 | Week 52
  Percentage of participants with clinical remission at Week 52 will be reported.
Cohorts 1 and 7: Percentage of Participants with Clinical Remission at Week 52 Evaluated by Ustekinumab Dose Bands | Week 52
  Percentage of participants with clinical remission at Week 52 evaluated by ustekinumab dose bands will be reported.
Cohorts 1 and 7: Percentage of Participants with Clinical Remission at Week 52 with No Corticosteroid Use | Week 52
  Percentage of participants with clinical remission at Week 52 with no corticosteroid use will be reported.
Cohorts 1 and 7: Percentage of Participants with Clinical Remission at Week 52 by PGA Score | Week 52
  Percentage of participants with clinical remission at Week 52 by Physician Global Assessment (PGA) score will be reported.
Cohorts 1 and 7: Change from Baseline in Height at Week 52 | Baseline and Week 52
  Change from baseline in height at Week 52 will be reported.
Cohorts 1 and 7: Change from Baseline in Weight at Week 52 | Baseline and Week 52
  Change from baseline in weight at Week 52 will be reported.
Cohorts 1 and 7: Change from Baseline in Body Mass Index (BMI) at Week 52 | Baseline and Week 52
  Change from baseline in BMI (measured with age and sex-specific z-scores) at Week 52 will be reported.
Cohorts 1 and 7: Percentage of Participants Who Achieve Endoscopic Remission with SEMA-CD Score of 0 or 1 at Week 52 | Week 52
  Percentage of participants who achieve endoscopic remission with simplified endoscopic mucosal assessment for Crohn's disease (SEMA-CD) score of 0 or 1 at Week 52 will be reported. Endoscopic remission is defined as SEMA-CD score of 0 or 1. SEMA-CD mucosal disease activity score is defined as inactive = 0; minimal = 1; mild = 2-4; moderate = 5-9, or severe = greater than or equal to (>=) 10.
Cohorts 1 and 7: Change from Baseline to Week 52 in Mucosal Disease Activity Measured with SEMA-CD Score | Baseline to Week 52
  Change from baseline to Week 52 in mucosal disease activity measured with SEMA-CD score will be reported. SEMA-CD mucosal disease activity score is defined as inactive = 0; minimal = 1; mild = 2-4; moderate = 5-9, or severe = greater than or equal to (>=) 10.
Cohorts 1 and 7: Percentage of Participants that Discontinued Ustekinumab Use Among Participants who Initiated Ustekinumab Therapy at Week 52 | Week 52
  Percentage of participants that discontinued ustekinumab use among participants who initiated ustekinumab therapy at Week 52 will be reported.
Cohorts 1 and 7: Percentage of Participants with Occurrence of Inflammatory Bowel Diseases (IBD)-related Hospitalizations Who had Initiated Ustekinumab Therapy | Up to Week 52
  Percentage of participants with occurrence of IBD-related hospitalizations who had initiated ustekinumab therapy will be reported.
Cohorts 1 and 7: Percentage of Participants with Occurrence of IBD-related Surgeries Who had Initiated Ustekinumab Therapy | Up to Week 52
  Percentage of participants with occurrence of IBD-related surgeries who had initiated ustekinumab therapy will be reported.
Cohorts 1 and 7: Percentage of Participants with Adverse Events of Special Interest (AESI) Who had Initiated Ustekinumab Therapy | Up to Week 52
  Percentage of participants with AESIs (example: malignancies, serious and opportunistic infection, anaphylaxis requiring discontinuation of ustekinumab) who had initiated ustekinumab therapy will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- ImproveCareNow, Inc., Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency